CLINICAL TRIAL: NCT02233868
Title: Brain Inflammation and Function in Alcoholism
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 140192; 14-AA-0192
Record Dates: First submitted 2014-09-06; First posted 2014-09-09 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-29

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: Imaging Studies; Alcohol Use Disorder (AUD); Inflammation
MeSH Terms: conditions — Alcoholism; Inflammation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I (Experimental): PET scan with [11C]PBR28 followed by PET scan with FDG and MRI.
  Interventions: Other: connectivity; Drug: neuroinflammation; Other: neurofunction
- Phase II (Experimental): After 3 weeks of abstinence or non-abstinence, PET scan with [11C]PBR28 followed by PET scan with FDG and MRI are repeated.
  Interventions: Other: connectivity; Drug: neuroinflammation; Other: neurofunction

INTERVENTIONS:
Other: connectivity — Magnetic resonance imaging (MRI) scans will be done to assess brain structure, functional reactivity and functional connectivity.
Drug: neuroinflammation — The use of [11C]PBR28 will allow us to assess for the first time in vivo if there is neuroinflammation in the brain of alcoholics. It will also allow us to assess if it recovers with alcohol detoxification.
Other: neurofunction — To assess regional brain glucose metabolism.

SUMMARY:
Background:

- Brain inflammation due to high alcohol intake may affect thinking, memory, and concentration. Researchers want to measure this using positron emission tomography (PET).

Objective:

- To study how excessive alcohol consumption affects brain function.

Eligibility:

* Adults 30-75 years old who are moderate or severe alcohol drinkers.
* Healthy volunteers.

Design:

* Participants will be screened with medical history, physical exam, interview, and blood and urine tests. Their breath will be tested for alcohol and recent smoking.
* Phase 1:
* Participants will stay in the hospital 3 days. They will have blood and heart tests and daily urine tests.
* A small plastic tube will be inserted by needle in each arm. One will go in a vein, the other in an artery.
* Participants will have 2 PET scans with 2 different radioactive compounds. Participants will lie on a bed that slides in and out of the scanner with a cap on their head.
* Participants will have magnetic resonance imaging (MRI) scans. Participants will lie in the scanner either resting with their eyes open or while performing an attention task.
* Participants will have tests of memory, attention, concentration, and thinking. They may answer questions, take tests, and perform simple actions.
* Phase 2 of the study will only be done if Phase 1 results show brain inflammation.
* Phase 2 will repeat Phase 1.
* For healthy volunteers, Phase 2 will begin 3 weeks after Phase 1.
* Other volunteers must not have alcohol for at least 3 weeks and stay in a hospital up to 4-6 weeks between Phase 1 and Phase 2. After Phase 2, they will have 5 follow-up calls over 3 months.

DETAILED DESCRIPTION:
The abuse of high doses of alcohol is associated with cognitive impairment that in extreme cases can result in dementia. However, the mechanisms underlying the neurotoxic effects of alcohol to the human brain are poorly understood. Here we test the hypothesis that alcohol-induced neuroinflammation contributes to its neurotoxic effects in humans

Objectives: The primary objectives in Phase I are to assess if there is inflammation in the brain of alcoholics and if present to determine if it recovers after at least 3 weeks of abstinence as compared between groups (alcoholic vs. healthy volunteers). Phase II objectives are to assess between group differences in inflammation in the brain of AUD subjects who either abstain from alcohol for at least 3 weeks or relapse (continue to drink alcohol) for at least 3 weeks. Secondary outcomes are to evaluate the functional consequences of inflammation as assessed by: regional brain glucose metabolism, functional brain activation to cognitive tasks, structural brain imaging, resting functional connectivity and neuropsychological tests.

Study population: Participants diagnosed with alcohol use disorder (AUD) as per DSM IV or DSM 5 AUD and healthy controls. Males and females ages 30-75 will be included.

Design: This study has two phases (phase I and II). The two phases can be done as inpatient (AUD subjects) or as outpatient (AUD and healthy controls) over a 2-3 day period. In phase I participants will undergo two positron emission tomography (PET) scans, one with [11C]PBR28 (marker of neuroinflammation) and one with 18FDG (marker of brain glucose metabolism) and magnetic resonance imaging (MRI) scans to assess brain structure, functional reactivity and functional connectivity. In parallel we will perform neuropsychological tests (NP). Phase II will include the same procedures as Phase I but it will be done at least 3 weeks later over a 2-3 day period only in AUD participants who successfully completed phase I who either abstained from alcohol or relapsed/continued to drink alcohol after Phase I. Relapsers would be eligible for Phase II if they continued to drink for at least 3 weeks prior scheduled imaging studies. We will complete Phase II studies on up to 24 additional AUD subjects (n=12 abstainers and n=12 relapsers) to assess whether [11C]PBR28 uptake recovers after abstinence. Since there are not much differences between test/retest studies in healthy volunteers in the literature [1], there is no need to complete Phase II studies in controls.

Outcome parameters: Main outcome measure is to assess if there is neuroinflammation with alcoholism and if it recovers with detoxification. Secondary outcome measures are: to assess if neuroinflammation is associated with markers of brain function, which include (1) regional brain glucose metabolism; (2) MRI based voxel-based morphometry (VBM) to assess cortical atrophy; (3) blood-oxygenation level-dependent (BOLD) activation to a cognitive task, (4) brain functional connectivity, (5) myo-inositol (mI) concentration, and (6) NP testing to assess cognitive performance, and to evaluate if neuroinflammation predicts relapse in AUD over a 3 month follow-up period.

[1] Collste K, Forsberg A, Varrone A, Amini N, Aeinehband S, Yakushev I, Halldin C, Farde L, Cervenka S. Test-retest reproducibility of [(11)C]PBR28 binding to TSPO in healthy control subjects. Eur J Nucl Med Mol Imaging. 2016 Jan;43(1):173-83. doi: 10.1007/s00259-015-3149-8. Epub 2015 Aug 22.

ELIGIBILITY:
-INCLUSION CRITERIA:

-All Participants

1. Between 30 and 75 years of age.
2. Ability to provide written informed consent as determined by physical examination and verbal communication. Capacity to consent will be determined by those giving the informed consent.
3. Females: Negative urine pregnancy test and not currently breastfeeding. Post-menopausal or surgically sterile (tubal ligation or hysterectomy); or not sexually active with a male partner and able to get pregnant; or documented agreement to use an effective form of birth control. Acceptable forms of contraception include: hormonal contraceptives (birth-control pills, injectable hormones, vaginal-ring hormones); IUD; diaphragm with spermicide; condom with spermicide.

   -Specific For AD Participants
4. DSM-IV diagnosis of alcohol dependence or alcohol abuse or DSM-5 diagnosis of moderate or severe alcohol use disorder (established through history and clinical exam). We include subjects that drink high doses of alcohol since alcohol's detrimental effects are greater with larger doses and particularly with binge drinking.
5. Participants seeking treatment for their AD as well as those not seeking treatment for their AD will be included.
6. Minimum 5 year history of heavy drinking (self-report).
7. Must consume at least 20 alcoholic drinks per week (male) or 15 per week (female) (self-report).
8. Must have had the last drinking episode (females 3 or more drinks; and males 4 or more drinks) within 1 week of baseline PET scan (self-report).
9. Alcohol specified as the preferred drug (self-report).

EXCLUSION CRITERIA:

* All Participants

  1. Unwilling or unable to refrain from use within 24 hours of scheduled study procedures: psychoactive medications or medication that may affect study results (e.g., analgesics [non narcotic], antibiotics (must finish course at least 24 hours prior to a scheduled procedure), antidiarrheal preparations, anti-inflammatory drugs (systemic corticosteroids are exclusionary), antinauseants, cough/cold preparations) (self-report, medical history). The following medications are allowable for entry on this study: analgesics (non-narcotic); antacids; antiasthma agents that are not systemic corticosteroids; antifungal agents for topical use; antihistamines (non-sedating); H2-Blockers/PPI (proton pump inhibitors); laxatives. The use of antihyperlipidemics and/or diuretics are permitted as long as they have been taken for at least 1 month before procedure visits and dose has been stabilized. The use of benzodiazepines such as alprazolam (( )Xanax), diazepam (( )Valium) and lorazepam (( )Ativan), will not exclude participants from this study.
  2. Current or past DSM-IV or DSM-5 diagnosis of a psychiatric disorder (other than alcohol in AD participants and nicotine/caffeine use disorders) that required hospitalization (any length), or chronic medication management (more than 4 weeks) and that could impact brain function at the time of the study as determined by history and clinical exam. The following chronically used medications are exclusionary from the study: analgesics containing narcotics; anorexics (sibuteramine); antianginal agents; antiarrhythmics; antiasthma agents that are systemic corticosteroids; antibiotics; anticholinergics; anticoagulants; anticonvulsants; antidepressants; antidiarrheal preparations; antifungal agents (systemic); antihistamines (sedating); antihypertensives; anti-inflammatory drugs (systemic); antineoplastics; antiobesity; antipsychotics; antivirals (except for treatment of HSV with agents without CNS activity, e.g. acyclovir, ganciclovir, famciclovir, valacyclovir); anxiolytics; cough/cold preparations (dextromethorphan preparations, pseudoephedrine); hormones (exceptions: thyroid hormone replacement, oral contraceptives, and estrogen replacement therapy); insulin; lithium; muscle relaxants; psychotropic drugs not otherwise specified (nos) including herbal products (no drugs with psychomotor effects or with anxiolytics, stimulant, antipsychotic, or sedative properties); sedatives/hypnotics. Note that nicotine and/or caffeine use will not exclude participants.
  3. Major medical problems that can permanently impact brain function (e.g., CNS, cardiovascular, metabolic, autoimmune, endocrine) as determined by history and clinical exam.
  4. Any clinically significant laboratory finding as determined during the screening procedures that could impact brain function or study procedures (evidenced from clinical laboratory results).
  5. Have had previous radiation exposure (from X-rays, PET scans, or other exposure) that with the exposure from this study, would exceed NIH annual research limits (self-report, medical history)
  6. Head trauma with loss of consciousness for more than 30 minutes (self-report, medical history);
  7. Positive test for alcohol on the day of the PET, the MRI or the NP tests (clinical laboratory results).
  8. Urine positive for psychoactive drugs (clinical laboratory results) on study days involving imaging (PET and MRI) and neuropsychological testing.
  9. Pregnant or breast feeding (self-report)
  10. History of coagulation disorder (clinical laboratory results, medical history)
  11. Have a history of allergic reaction to lidocaine (self-report, medical history)
  12. Presence of ferromagnetic objects in the body that are contraindicated for MRI of the head, fear of enclosed spaces, or other standard contraindication to MRI (self-report checklist).
  13. Cannot lie comfortably flat on your back for up to 2 hours in the PET and MRI scanners (self-report).
  14. Body weight > 250 kg. The MR scanner bed is tested to a weight limit of 250 kg (~550 lbs).
  15. Have a positive HIV test (clinical laboratory results, medical history).
  16. Homozygosity for the rs6971 polymorphism on TSPO that results in LB (Owen et al 2011) (genotyping results).
  17. NIH employees who meet criteria as AD subjects. Although we will include NIH employees as healthy volunteers, study investigators and their superiors, subordinates and immediate family members (adults children, spouses, parents, siblings) will be excluded.

      EXCLUSION CRITERIA SPECIFIC FOR CONTROL PARTICIPANTS:
* Consumption of moderate to high levels of alcohol. That includes if female, currently (within past 6 months) consuming more than 2 drinks on a given episode and if male, consuming more than 3 drinks on a given episode; and/or consuming if female, more than a total of 7 drinks a week or if male, more than 10 drinks a week (self-report).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-02-19 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
To determine if there is neuroinflammation in the brain. | end of study
  To assess if there is neuroinflammation detected in the brain of alcoholics subjects as measured with [11C]PBR28 as compared to healthy controls and if it recovers with at least 3 weeks of abstinence.
To assess inflammation in brain. | end of study
  To assess if there is inflammation detected in the brain of alcoholics subjects as measured with [11C]PBR28 as compared to healthy controls.
To assess between group differences in inflammation in the brain of AUD subjects in Phase II who either abstain from alcohol for at least 3 weeks or relapse (continue to drink alcohol) for at least 3 weeks. | end of study
  We want to see whether [11C]PBR28 uptake in the brain reflects levels similar to controls after at least 3 weeks of alcohol abstinence.

SECONDARY OUTCOMES:
To assess the impact of neuroinflammation on brain function (assessed with PET and 18FDG and with MRI for fMRI with task activation and for functional connectivity). | end of study
  to assess if neuroinflammation is associated with markers of brain function and to evaluate if neuroinflammation predicts relapse in AUD over a 3 month follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Dardo G Tomasi, Ph.D., Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Data is analyzed by subject group and not on an individual basis.

REFERENCES:
- [Derived] Paul S, Gallagher E, Liow JS, Mabins S, Henry K, Zoghbi SS, Gunn RN, Kreisl WC, Richards EM, Zanotti-Fregonara P, Morse CL, Hong J, Kowalski A, Pike VW, Innis RB, Fujita M. Building a database for brain 18 kDa translocator protein imaged using [11C]PBR28 in healthy subjects. J Cereb Blood Flow Metab. 2019 Jun;39(6):1138-1147. doi: 10.1177/0271678X18771250. Epub 2018 May 11. PMID 29749279
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-AA-0192.html